CLINICAL TRIAL: NCT00733213
Title: Depiction of Prostate Cancer Treatment Alternatives in Greece
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Dr Pontikis Panagiotis, MD Medical and Regulatory Affairs Director, AstraZeneca, SA Greece
Other Study IDs: NIS-OGR-DUM-2007/1
Record Dates: First submitted 2008-08-08; First posted 2008-08-12 (Estimated); Last update posted 2009-10-14 (Estimated); Status verified 2009-10

CONDITIONS: Locally Advanced or Metastatic Prostate Cancer.
Keywords: Prostate Cancer, Treatment alternatives, Metastasis
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A retrospective, registry analysis of the socio-economic and demographic characteristics of patients suffering from locally advanced or metastatic prostate cancer, as well as the depiction of the therapeutic algorithms followed in the Greek clinical practice.

* Target Group: Patients with locally advanced or metastatic prostate cancer.
* The first 10 consecutive patients records that meet the entry criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Locally advanced or Metastatic Prostate Cancer after 2002.
* Patients that received Hormonal therapy.

Exclusion Criteria:

* Males that are aged less than 18 years

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Target Group: Patients diagnosed with Locally advanced or Metastatic Prostate Cancer
Sampling Method: Probability Sample
Enrollment: 310 (Estimated)
Dates: Start 2008-01; Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Percentage of patients treated by each treatment alternative. | Between 2002 - 2008

SECONDARY OUTCOMES:
To depict sociodemographic characteristics and comorbidities. | Between 2002 - 2008

CONTACTS AND LOCATIONS:
Overall Officials: Panagiotis Pontikis, MD, Study Director — AstraZeneca Greece
Locations (4):
- Greece (4):
  - Research Site, Athens
  - Research Site, Karditsa
  - Research Site, Serres
  - Research Site, Xsanthi